CLINICAL TRIAL: NCT04366739
Title: Repurposing of Chlorpromazine in Covid-19 Treatment
Acronym: reCoVery
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: No favourable opinion obtained from the Ethics Committee
Sponsor: Centre Hospitalier St Anne (Other)
Collaborators: Hôpital Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D20-P016
Record Dates: First submitted 2020-04-24; First posted 2020-04-29 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2020-04

CONDITIONS: COVID-19
Keywords: COVID-19; Chlorpromazine
MeSH Terms: conditions — COVID-19 | interventions — Chlorpromazine; Standard of Care

STUDY DESIGN:
Intervention Model Description: Allocation: Randomized Intervention Model: Parallel Assignment
  Intervention Model Description:
  reCoVery is a multi-center, randomized, single-blind, standard care-controlled (1:1) pilot clinical study to explore the efficacy and safety of chlorpromazine (CPZ) in the treatment of adult subjects with COVID-19-moderate type (WHO-OSCI 3-5).
Who Masked: Outcomes Assessor
Masking Description: The evaluator of the primary endpoint and secondary endpoints relating to the clinical efficacy of CPZ and the evaluator of the biological and radiological effects of the CPZ will be maintained blindly throughout their duration of inclusion. This evaluator will collect clinical data, biological data, and imaging data without knowing the drug treatments delivered to patients.
  The radiologists responsible for calculating the parenchymal damage score on the thoracic CT scan will be blind to the patient delivered drugs.
  The biologists responsible for carrying out the analyzes on the biobank will be blind to the patient delivered drugs.
  The biostatistician responsible for statistical study analysis will be kept blind to the drugs delivered to the subjects.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CHLORPROMAZINE (CPZ) (Experimental): Standard of Care (SOC) plus CHLORPROMAZINE (CPZ)
  Interventions: Drug: CHLORPROMAZINE (CPZ); Combination Product: Standard of Care (SOC)
- standard of care (SOC) (Active Comparator): In the absence of a reference treatment in COVID-19, the "standard of care" (SOC) is the comparator arm
  Interventions: Combination Product: Standard of Care (SOC)

INTERVENTIONS:
Drug: CHLORPROMAZINE (CPZ) — Drug List 1, AMM obtained in 1952, AMM 3400930571187 1952/90, RCP revised 22/08/2019 Administration: oral route, if the clinical condition requires it, intravenous administration.
  Initial dosage: 75 mg per day orally (or 37.5 mg per day orally in subjects 75 years of age or older).
  Then: titration up to the maximum tolerated dose, with a minimum of 12.5 mg and a maximum of 300 mg per day by the oral administration (or 600 mg per day by the oral in certain exceptional cases which also correspond to the CPM CPM marketing authorization indications); or from 6.25 to 150 mg per day intravenously.
  Duration of treatment: until healing criteria are obtained (≥ 8 days from the onset of COVID-19 symptoms AND ≥ 48 hours of apyrexia and absence of dyspnea) or 21 days maximum
  Arms: CHLORPROMAZINE (CPZ)
Combination Product: Standard of Care (SOC) — In the absence of a reference treatment in COVID-19, the "standard of care" (SOC) is the comparison arm

SUMMARY:
This study evaluates the effects of the addition of chlorpromazine to the standard therapeutic protocol in COVID-19 patients hospitalized for respiratory symptom management (score 3-5 WHO Ordinal Scale for Clinical Improvement).

DETAILED DESCRIPTION:
This study evaluates the effects of the addition of chlorpromazine to the standard therapeutic protocol in COVID 19 patients hospitalized for respiratory symptom management (score 3-5 WHO Ordinal Scale for Clinical Improvement).

The investigators have observed in GHU-Paris psychiatry Hospital units (140 beds), significantly lower prevalence of symptomatic and severe forms of COVID-19 in patients (3%) than in the health workers operating in the same facilities (19% of nurses and 18% of physicians). COVID-psychiatry units report similar feedback in France, Spain, and Italy. One hypothesis could be that psychotropic drugs have a protective action on COVID-19 and protect patients from symptomatic and virulent forms of COVID-19.

This hypothesis is consistent with research studies that have shown that several psychotropic drugs inhibit in vitro viral replication of the coronaviruses MERS-CoV and SARS-CoV-1. The SARS-CoV-2 has many characteristics in common with the coronavirus family and has phylogenetic similarities to the SARS-CoV-1 engaged in the 2002-2003 outbreak. It is, therefore, possible that one or more psychotropic drugs having demonstrated efficacy against MERS-CoV and SARS-CoV-1 also have anti-SARS-CoV-2 antiviral activity.

The current global epidemic of COVID-19, with a high number of deaths in many countries, makes it urgent to search drugs potentially useful to reduce the severity and lethality of the infection. Drug repositioning represents a possible alternative to the news medicines discovery. This strategy makes it possible to eliminate many stages of development; it makes it possible to deploy a therapy whose side effects are known and which physicians already well know how to handle.

To confirm the hypothesis of the antiviral action of chlorpromazine on SARS-CoV-2, a preclinical in vitro experiment began in April 2020 at the level III high-security biological laboratory at the Pasteur Institute (in collaboration with the GHU PARIS Psychiatry & Neurosciences). The first results are encouraging and show a marked antiviral effect of chlorpromazine on SARS-CoV-2. Technical replicas are underway to validate these preliminary results.

By integrating all these evidence, the investigators hypothesize that chlorpromazine could decrease the unfavorable evolution of COVID-19 infection when administered at the onset of respiratory signs.

ELIGIBILITY:
Inclusion Criteria:

* Biological and/or radiological diagnosis of COVID-19 infection
* WHO-OSCI at 3, 4 or 5 at the time of inclusion
* Benefiting from a social security scheme
* Voluntarily participating in the clinical study; fully understanding and being fully informed of the study and having signed the Informed Consent Form (ICF); willingness and capability to complete all the study procedures

Exclusion Criteria:

* Treatment with chlorpromazine (CPZ) the month preceding the inclusion visit
* Contraindication to the CPZ:
* Hypersensitivity to the active substance or any of the excipients
* Risk of glaucoma by closing the angle.
* Risk of urinary retention linked to urethroprostatic disorders.
* History of agranulocytosis
* Association with dopaminergic outside Parkinson's (cabergoline, quinagolide), citalopram, escitalopram, domperidone, hydroxyzine, and piperaquine
* Wheat allergy
* Risk of QT prolongation and occurrence of severe ventricular rhythm disorders: the existence of bradycardia, hypokalaemia, long congenital or acquired QT
* History of ischemic stroke
* Treatment with chloroquine or hydroxychloroquine during the inclusion visit or the previous month
* Need for mechanical ventilation linked to COVID-19, during the inclusion visit or the last month
* In the opinion of the clinical team, imminent progression to death within the next 24 hours regardless of treatment
* Psychiatric care under duress
* Protected adults, persons under the protection of justice
* Pregnant or lactating woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-04-29 (Estimated); Primary Completion 2020-08-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Time To Response (TTR) | 28 days
  The primary endpoint is the time to response (TTR) in days, from randomization to 28th day. By response to treatment is meant the reduction of at least one severity level on the World Health Organization Ordinal Scale for Clinical Improvement (WHO-OSCI)
  The WHO-OSCI is an ordinal scale of 9 severity levels (from 0 to 8) for COVID-19. This scale was established by the WHO, which recommends its use for any therapeutic study on COVID-19.
  This will be a continuous outcome defined by the amount of time between randomization to the first response. This will be treated as a time-to-event with possible censoring.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 28 days from randomization
  Response rate regarding the World Health Organization Ordinal Scale for Clinical Improvement (WHO-OSCI).
  This will be a binary outcome defined by clinical conditions improvement assessment from randomization to 28th Day, by the response to treatment is meant the reduction of at least one severity level on the World Health Organization Ordinal Scale for Clinical Improvement (WHO-OSCI).
All-cause mortality | 28 days after randomization
  All-cause mortality rates at Day 28th after randomization
Duration in days required for hospital discharge | 28 days after randomization
  This will be a continuous outcome defined by the amount of time in days between randomization and the hospital discharge
Duration in days required for National Early Warning Score ≤ 2 maintained 24 hours | 28 days after randomization
  This will be a continuous outcome defined by the amount of time in days between randomization and National Early Warning Score ≤ 2 maintained for almost 24 hours
  The National Early Warning Score (NEWS) is a score used in the ICU to evaluate the overall severity of the clinical condition of a patient.
Number of days without oxygen therapy | 28 days after randomization
  This will be a continuous outcome defined by the amount of time in days without oxygen therapy
Incidence of oxygen use, NIV or high flow oxygen therapy | 28 days after randomization
  Number of clinical conditions that need a prescription for Oxygen therapy, NIV or high flow oxygen therapy
Duration in days of oxygen prescription, NIV or high flow oxygen therapy | 28 days after randomization
  This will be a continuous outcome defined by the amount of time in days with oxygen therapy, NIV, or high flow oxygen therapy.
Biochemical response: rate of patients positive for SARS-CoV-2 PCR on a nasopharyngeal sample | day 7 from randomization
  Rate of patients positive for SARS-CoV-2 PCR on a nasopharyngeal sample (biobank sample) (day 7) This will be a binary outcome defined by positive or negative results at SARS-CoV-2 PCR on a nasopharyngeal sample
Biochemical response: viral load of SARS-CoV-2 on a nasopharyngeal sample | day 7 from randomization
  This will be a quantitative variable. Biobank sample at day 7
Biochemical response: serum viral load of SARS-CoV-2 | day: 3,5,7,14,21,28
  This will be a quantitative variable. Biobank blood sample at D3, D5, D7 then, if hospitalization continues blood sample at D14, D21, and D28
Biochemical response: C-reactive protein (CRP) | day: 3,5,7,14,21,28
  This will be a quantitative variable. Biobank blood sample at D3, D5, D7 then, if hospitalization continues blood sample at D14, D21, and D28
Biochemical response: blood test for lymphocytes (lymphopenia) | day: 3,5,7,14,21,28
  This will be a quantitative variable. Biobank blood sample at D3, D5, D7 then, if hospitalization continues blood sample at D14, D21, and D28
Parenchymal involvement (chest CT) | day 7
  Extension score of parenchymal involvement in thoracic computed tomography (CT) (D7)
Define the optimal dose of CPZ and its tolerance: rates of serious adverse events | 28 days
  Rates of serious adverse events
Define the optimal dose of CPZ and its tolerance: rates of non-serious side effects | 28 days
  Rates of non-serious side effects
Define the optimal dose of CPZ and its tolerance: anxiety assessment on Global Anxiety - Visual Analog Scale (GA-VAS) | 28 days
  Global Anxiety - Visual Analog Scale (GA-VAS) is a scale for the assessment of anxiety. The 100 mm GA-VAS varies from minimum (not at all anxious) to maximum (Extremely anxious).
  This will be a quantitative variable, the distance from the left edge of the line to the mark placed by the patient is measured to the nearest millimeter and used in analyses as the patient's GA-VAS score.
Define the optimal dose of CPZ and its tolerance: Rates of drug discontinuation | 28 days
  Rates of drug discontinuation in all causes under study
Define the optimal dose of CPZ and its tolerance: biological anomalies | day: 3,5,7,14,21,28
  NFS, TP TCA, blood ionogram and hepatic check-up, glycemia. This will be a quantitative variable. Biobank blood sample at D3, D5, D7 then, if hospitalization continues blood sample at D14, D21, and D28
Define the optimal dose of CPZ and its tolerance: ECG abnormalities | day: 3,5,7,14,21,28
  Rate of patients with ECG abnormalities at D3, D5, D7 then, if hospitalization continues blood sample at D14, D21, and D28
Define the optimal dose of CPZ and its tolerance: plasma CPK assessment | day: 3,5,7,14,21,28
  plasma CPK assessment at D3, D5, D7 then, if hospitalization continues blood sample at D14, D21, and D28
Define the optimal dose of CPZ and its tolerance:plasma CPZ assessment | day: 3,5,7,14,21,28
  Plasma CPZ assessment at D3, D5, D7 then, if hospitalization continues blood sample at D14, D21, and D28
Define the optimal dose of CPZ and its tolerance: CPZ dose administered | 28 days
  CPZ dosages administered

OTHER OUTCOMES:
Evaluate the biological parameters to treatment response (biobank constitution for carrying out cytokine assays, lymphocyte profiles in flow cytometry and additional explorations according to the evolution of knowledge on COVID-19) | day: 1, 3,5,7,14,21,28
  Biobank by blood samples of 20 ml per patient (on D1, D3, D5, D7, then, if continued hospitalization at D14, D21, D28) allowing, in addition to viral markers:Cytokine and lymphocyte profile assays in flow cytometry: IL-2, IL-6, IL-7, IL-10, GCSF, IP10, MCP1, M1P1A and TNF-alfa, FACs CD3, CD4, CD8, CD38

CONTACTS AND LOCATIONS:
Overall Officials: Marion Plaze, MD, PHD, Principal Investigator — Service Hospitalo-Universitaire - GHU PARIS Psychiatrie & Neurosciences
Locations (1):
- Centre Hospitalier Sainte-Anne, Paris, France

REFERENCES:
- [Background] Blanchard E, Belouzard S, Goueslain L, Wakita T, Dubuisson J, Wychowski C, Rouille Y. Hepatitis C virus entry depends on clathrin-mediated endocytosis. J Virol. 2006 Jul;80(14):6964-72. doi: 10.1128/JVI.00024-06. PMID 16809302
- [Background] Burkard C, Verheije MH, Wicht O, van Kasteren SI, van Kuppeveld FJ, Haagmans BL, Pelkmans L, Rottier PJ, Bosch BJ, de Haan CA. Coronavirus cell entry occurs through the endo-/lysosomal pathway in a proteolysis-dependent manner. PLoS Pathog. 2014 Nov 6;10(11):e1004502. doi: 10.1371/journal.ppat.1004502. eCollection 2014 Nov. PMID 25375324
- [Background] Calsina-Berna A, Garcia-Gomez G, Gonzalez-Barboteo J, Porta-Sales J. Treatment of chronic hiccups in cancer patients: a systematic review. J Palliat Med. 2012 Oct;15(10):1142-50. doi: 10.1089/jpm.2012.0087. Epub 2012 Aug 14. No abstract available. PMID 22891647
- [Background] Chu VC, McElroy LJ, Bauman BE, Whittaker GR. Fluorescence dequenching assays of coronavirus fusion. Adv Exp Med Biol. 2006;581:241-6. doi: 10.1007/978-0-387-33012-9_40. No abstract available. PMID 17037536
- [Background] Cong Y, Hart BJ, Gross R, Zhou H, Frieman M, Bollinger L, Wada J, Hensley LE, Jahrling PB, Dyall J, Holbrook MR. MERS-CoV pathogenesis and antiviral efficacy of licensed drugs in human monocyte-derived antigen-presenting cells. PLoS One. 2018 Mar 22;13(3):e0194868. doi: 10.1371/journal.pone.0194868. eCollection 2018. PMID 29566060
- [Background] Daniel JA, Chau N, Abdel-Hamid MK, Hu L, von Kleist L, Whiting A, Krishnan S, Maamary P, Joseph SR, Simpson F, Haucke V, McCluskey A, Robinson PJ. Phenothiazine-derived antipsychotic drugs inhibit dynamin and clathrin-mediated endocytosis. Traffic. 2015 Jun;16(6):635-54. doi: 10.1111/tra.12272. Epub 2015 Apr 9. PMID 25693808
- [Background] de Wilde AH, Jochmans D, Posthuma CC, Zevenhoven-Dobbe JC, van Nieuwkoop S, Bestebroer TM, van den Hoogen BG, Neyts J, Snijder EJ. Screening of an FDA-approved compound library identifies four small-molecule inhibitors of Middle East respiratory syndrome coronavirus replication in cell culture. Antimicrob Agents Chemother. 2014 Aug;58(8):4875-84. doi: 10.1128/AAC.03011-14. Epub 2014 May 19. PMID 24841269
- [Background] Dyall J, Coleman CM, Hart BJ, Venkataraman T, Holbrook MR, Kindrachuk J, Johnson RF, Olinger GG Jr, Jahrling PB, Laidlaw M, Johansen LM, Lear-Rooney CM, Glass PJ, Hensley LE, Frieman MB. Repurposing of clinically developed drugs for treatment of Middle East respiratory syndrome coronavirus infection. Antimicrob Agents Chemother. 2014 Aug;58(8):4885-93. doi: 10.1128/AAC.03036-14. Epub 2014 May 19. PMID 24841273
- [Background] Marmura MJ, Silberstein SD, Schwedt TJ. The acute treatment of migraine in adults: the american headache society evidence assessment of migraine pharmacotherapies. Headache. 2015 Jan;55(1):3-20. doi: 10.1111/head.12499. PMID 25600718
- [Background] Pohjala L, Utt A, Varjak M, Lulla A, Merits A, Ahola T, Tammela P. Inhibitors of alphavirus entry and replication identified with a stable Chikungunya replicon cell line and virus-based assays. PLoS One. 2011;6(12):e28923. doi: 10.1371/journal.pone.0028923. Epub 2011 Dec 19. PMID 22205980
- [Background] Pu Y, Zhang X. Mouse hepatitis virus type 2 enters cells through a clathrin-mediated endocytic pathway independent of Eps15. J Virol. 2008 Aug;82(16):8112-23. doi: 10.1128/JVI.00837-08. Epub 2008 Jun 11. PMID 18550663
- [Background] Verity R, Okell LC, Dorigatti I, Winskill P, Whittaker C, Imai N, Cuomo-Dannenburg G, Thompson H, Walker PGT, Fu H, Dighe A, Griffin JT, Baguelin M, Bhatia S, Boonyasiri A, Cori A, Cucunuba Z, FitzJohn R, Gaythorpe K, Green W, Hamlet A, Hinsley W, Laydon D, Nedjati-Gilani G, Riley S, van Elsland S, Volz E, Wang H, Wang Y, Xi X, Donnelly CA, Ghani AC, Ferguson NM. Estimates of the severity of coronavirus disease 2019: a model-based analysis. Lancet Infect Dis. 2020 Jun;20(6):669-677. doi: 10.1016/S1473-3099(20)30243-7. Epub 2020 Mar 30. PMID 32240634
- [Background] Wang D, Hu B, Hu C, Zhu F, Liu X, Zhang J, Wang B, Xiang H, Cheng Z, Xiong Y, Zhao Y, Li Y, Wang X, Peng Z. Clinical Characteristics of 138 Hospitalized Patients With 2019 Novel Coronavirus-Infected Pneumonia in Wuhan, China. JAMA. 2020 Mar 17;323(11):1061-1069. doi: 10.1001/jama.2020.1585. PMID 32031570
- [Background] Wang LH, Rothberg KG, Anderson RG. Mis-assembly of clathrin lattices on endosomes reveals a regulatory switch for coated pit formation. J Cell Biol. 1993 Dec;123(5):1107-17. doi: 10.1083/jcb.123.5.1107. PMID 8245121
- [Background] Weinman D, Nicastro O, Akala O, Friedman BW. Parenteral treatment of episodic tension-type headache: a systematic review. Headache. 2014 Feb;54(2):260-8. doi: 10.1111/head.12287. Epub 2014 Jan 16. PMID 24433525
- [Background] Zhu N, Zhang D, Wang W, Li X, Yang B, Song J, Zhao X, Huang B, Shi W, Lu R, Niu P, Zhan F, Ma X, Wang D, Xu W, Wu G, Gao GF, Tan W; China Novel Coronavirus Investigating and Research Team. A Novel Coronavirus from Patients with Pneumonia in China, 2019. N Engl J Med. 2020 Feb 20;382(8):727-733. doi: 10.1056/NEJMoa2001017. Epub 2020 Jan 24. PMID 31978945